CLINICAL TRIAL: NCT00266448
Title: The Value of Whole Body Washing With Chlorhexidine for the Eradication of MRSA - a Randomized, Placebo-Controlled, Double-Blinded Clinical Trial
Brief Title: Whole Body Washing With Chlorhexidine for the Eradication of MRSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 94/2000; Projekt-Nr. 384/2000
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2004-04

CONDITIONS: MRSA-Colonization
Keywords: MRSA; eradication; chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine solution 4%

SUMMARY:
The purpose of this study is to determine whether whole body washing with chlorhexidine in combination with mupirocine nasal ointment is effective in the eradication of meticillin-resistant Staphylococcus aureus (MRSA).

DETAILED DESCRIPTION:
The number and rate of infections due to meticillin-resistant Staphylococcus aureus (MRSA)is increasing world wide. Patients who are colonized with MRSA are the main source for further distribution. In addition colonization with MRSA is a precondition for infection.

Whole body washing with antiseptic solutions as part of eradication strategies for MRSA has been widely used. However, there is insufficient evidence to support use of topical antimicrobial therapy for eradicating of MRSA because treatment with antiseptic solution has never been compared to placebo.

Comparison: The efficacy of whole body washing in the control of MRSA was studied in a randomized, placebo-controlled, double-blinded clinical trial. The study treatment consisted of five days of whole body washing either with 4% chlorhexidine solution (verum) or with placebo. All patients received mupirocin nasal ointment and chlorhexidine mouth rinse. The outcome was evaluated 3, 4, 5, 9 and 30 days after treatment by swabs taken from several body site.

ELIGIBILITY:
Inclusion Criteria:

* persons who are colonized with MRSA, i.e. one or more cultures from any body site yielded MRSA

Exclusion Criteria:

* ongoing systemic or local antimicrobial treatment directed against MRSA
* hypersensitivity to mupirocin or chlorhexidine
* pregnancy
* previous enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-01; Study Completion 2004-04

PRIMARY OUTCOMES:
efficacy of a whole body treatment with chlorhexidine in eradicating overall MRSA carriage

SECONDARY OUTCOMES:
development of MRSA infection
tolerance to the antiseptic whole body treatment

CONTACTS AND LOCATIONS:
Overall Officials: Constanze Wendt, MD, MSc, Principal Investigator — Hygiene-Institut University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Wendt C, Schinke S, Wurttemberger M, Oberdorfer K, Bock-Hensley O, von Baum H. Value of whole-body washing with chlorhexidine for the eradication of methicillin-resistant Staphylococcus aureus: a randomized, placebo-controlled, double-blind clinical trial. Infect Control Hosp Epidemiol. 2007 Sep;28(9):1036-43. doi: 10.1086/519929. Epub 2007 Jul 3. PMID 17932823